CLINICAL TRIAL: NCT04474418
Title: Be-PART: Berlin Psychometric Characterization of Patients With Cardiac ARrhyThmias
Brief Title: Psychometric Characterization of Patients With Cardiac Arrhythmias
Acronym: Be-PART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Dr. Jens Plag, MD, Charite University, Berlin, Germany
Other Study IDs: EA2/211/17
Record Dates: First submitted 2020-07-02; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Cardiac Arrhythmia; Anxiety; Personality; Psychological Stress; Depression
Keywords: cardiac arrhythmia, personality, psychological symptoms
MeSH Terms: conditions — Arrhythmias, Cardiac; Anxiety Disorders; Stress, Psychological; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the influence of different psychological parameters (e.g. depression, anxiety, personality traits, resilience, tolerance of uncertainty or heart beat perception) on treatment outcome and quality of life in patients with cardiac arrythmias.

DETAILED DESCRIPTION:
This longitudinal observational study examines patients with cardiac arrhythmia (such as atrial fibrillation or atrial flutter) who are undergoing a conventional standard therapy in the Department of Cardiology of the Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin. To examine the impact of psychological symptoms such as anxiety, depression, resilience and risk factors (e.g. neuroticism) on cardiac treatment outcomes, patients are evaluated with a standardized psychological assessment including established questionnaires. The baseline observation is performed before the standard treatment of the arrhythmia (e.g. pharmacological treatment or electrophysiological methods). Follow-up observations are made 3 and 6 month after the cardiological intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority (min. 18 years old)
* no severe cognitive dysfunction
* diagnosed cardiac arrhythmias
* reason of admission is the treatment of cardiac arrhythmia

Exclusion Criteria:

* medium to severe cognitive dysfunction
* doubt on capacity to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with cardiac arrythmias without any signs of medium or severe cognitive dysfunction.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) - Change from Baseline at 6 months | From Baseline at 6 months (Follow-up) after standard therapy
  BDI is a questionnaire measuring depression

SECONDARY OUTCOMES:
NEO-FFI personality inventory | Only at baseline
  personality inventory measuring neuroticism, extraversion, openness to experience, agreeableness, conscientiousness
Electrocardiography (ECG) - Change from Baseline at 6 months | From Baseline at 6 months (Follow-up) after standard therapy
  measuring heart activity and signs of cardiac arrhythmias
Heart beat Counting Task by Schandry | Baseline
  Assessment of patients heart beat perception
Angstkontrollfragebogen (AKF) - Baseline | Baseline before standard therapy
  AKF is the German Version of the Anxiety Control Questionnaire
Angstkontrollfragebogen (AKF) - 3 months after standard therapy | 3 months after standard therapy
  AKF is the German Version of the Anxiety Control Questionnaire
Angstkontrollfragebogen (AKF) - 6 months after standard therapy | 6 months after standard therapy
  AKF is the German Version of the Anxiety Control Questionnaire
Anxiety Sensitivity Index (ASI) - Baseline Anxiety Sensitivity Index (ASI) | Baseline
  ASI is a Questionnaire measuring anxiety sensitivity
Anxiety Sensitivity Index (ASI) - 3 months after standard therapy Anxiety Sensitivity Index (ASI) | 3 months after standard therapy
  ASI is a Questionnaire measuring anxiety sensitivity
Anxiety Sensitivity Index (ASI) - 6 months after standard therapy Anxiety Sensitivity Index (ASI) | 6 months after standard therapy
  ASI is a Questionnaire measuring anxiety sensitivity
Beck Anxiety Inventory (BAI) - Change from Baseline at 6 months | From Baseline at 6 months (Follow-up) after standard therapy
  BAI is a questionnaire measuring anxiety
Heart rate variability - Baseline | Baseline before standard therapy
  heart rate variability is a non-invasive method to measure autonomic nervous system function
Heart rate variability - 3 months after standard therapy | 3 months after standard therapy
  heart rate variability is a non-invasive method to measure autonomic nervous system function
Heart rate variability - 6 months after standard therapy | 6 months after Standardtherapie
  heart rate variability is a non-invasive method to measure autonomic nervous system function
Resilienzskala (RS-13) - Baseline | Baseline
  Questionnaire to measure resilience
Resilienzskala (RS-13) - 3 months after standard therapy | 3 months after standard therapy
  Questionnaire to measure resilience
Resilienzskala (RS-13) - 6 months after standard therapy | 6 months after standard therapy
  Questionnaire to measure resilience
Skala zur allgemeinen Selbstwirksamkeitserwartung (SWE) - Baseline | Baseline
  Questionnaire to measure self-efficacy
Skala zur allgemeinen Selbstwirksamkeitserwartung (SWE) - 3 months after standard therapy | 3 months after standard therapy
  Questionnaire to measure self-efficacy
Skala zur allgemeinen Selbstwirksamkeitserwartung (SWE) - 6 months after standard therapy | 6 months after standard therapy
  Questionnaire to measure self-efficacy
ICD-10-Symptom-Rating (ISR) - Change from Baseline at 6 months | From Baseline at 6 months after standard therapy
  Questionnaire to assess symptoms of psychiatric disorders
Perceived Stress Questionnaire (PSQ) - Change from Baseline at 6 months | From Baseline at 6 months after standard therapy
  Questionnaire to measure psychological stress perception
Body Sensations Questionnaire (BSQ) - Change from Baseline at 6 months | From Baseline at 6 months after standard therapy
  Questionnaire to measure body sensations related to anxiety
Herzangstfragebogen (HAF-17) - Change from Baseline at 6 | From Baseline at 6 months after standard therapy
  Questionnaire to measure anxiety with respect to cardiac symptoms
Fragebogen zu Akzeptanz und Handeln II (FAH-II) - Change from Baseline at 6 months | From Baseline at 6 months after standard therapy
  Questionnaire to measure psychological flexibility
Euroquol EQ-5D-3L - Change from Baseline at 6 | From Baseline at 6 months after standard therapy
  Questionnaire to measure quality of life
Unsicherheitsintoleranzfragebogen (UI-18) | Baseline
  Questionnaire to measure tolerance to uncertainty

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided